CLINICAL TRIAL: NCT01698489
Title: The Very Large Database of Lipids (VLDL): A Clinical Laboratory Big Data Project
Brief Title: The Very Large Database of Lipids
Acronym: VLDL
Status: Active, not recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: VAP Diagnostics Lab (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB00520613-2; NCT07169266 (obsolete NCT alias)
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Lipid Disorders and Lipid Measurement
MeSH Terms: conditions — Lipid Metabolism Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Closer examination of granular lipid data in a large population offers numerous opportunities to generate new knowledge, ranging from studies examining concordance between commonly used lipid parameters to phenotypic characterization of rare or extreme disorders of lipid metabolism, opening possibilities to better personalize future treatment of abnormal blood lipids.

STUDY POPULATION:

The Very Large Database of Lipids (VLDL) includes adults and children who were clinically referred for a Vertical Auto Profile (VAP). Patient samples originated predominantly from outpatient primary care clinics in the U.S. (85%), along with specialty clinics and inpatient settings.

LIPID MEASUREMENTS:

The VAP test (VAP Diagnostics Lab, Birmingham, Alabama, USA) directly measures cholesterol concentrations of low density lipoprotein, very low density lipoprotein, intermediate density lipoprotein, high density lipoprotein, their subfractions, and lipoprotein(a). Triglycerides in the database are directly measured using the Abbott ARCHITECT C-8000 system (Abbott Park, Illinois, USA). Lipid distributions in the database closely match those from the population-representative National Health and Nutrition Examination Survey (NHANES).

STUDY PROCEDURES:

This database was investigator-initiated. Only de-identified data reach the investigational site. The master database is housed at The Johns Hopkins Hospital in Baltimore, Maryland, and maintained by Drs. Jones and Martin. The current database (2nd harvest) includes 5,051,467 patients whose laboratory samples were collected from October 1, 2015 and June 30, 2019. Only electronic data, and not blood samples, are sent to Hopkins. The academic investigators have unrestricted access to study data, take responsibility for the accuracy of analyses, and have authority over manuscript preparation and submission.

VARIABLES:

The variables currently in the VLDL database are testing date, age, sex, fasting/nonfasting, and components of the VAP test. From these primary variables, many additional variables were derived for inclusion in the master database. Other analytes measured by validated assays in subsets of the VLDL database include apolipoprotein B (apoB), apolipoprotein A1 (apoAI), high-sensitivity C-reactive protein (hsCRP), homocysteine, uric acid, insulin, hemoglobin A1c, 25-hydroxy vitamin D, cystatin C, lipoprotein-associated phosphatase (Lp-PLA2), thyroid stimulating hormone (TSH), free T3 and T4, pro-brain natriuretic peptide (pBNP), direct bilirubin, creatine phosphokinase (CPK), creatinine and other components of the comprehensive metabolic panel, magnesium, and phosphate.

ELIGIBILITY:
Patients with age and lipid data are included in the master database. Eligibility criteria are specific to each individual study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients clinically referred for VAP density gradient ultracentrifugation.
Sampling Method: Non-Probability Sample
Enrollment: 5051467 (Actual)
Dates: Start 2006-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Low-density lipoprotein cholesterol level | 4 years
  Low-density lipoprotein cholesterol levels measured in milligrams per deciliter.

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Jones, MD, Study Director — Johns Hopkins University; Seth S Martin, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] Martin SS, Blaha MJ, Toth PP, Joshi PH, McEvoy JW, Ahmed HM, Elshazly MB, Swiger KJ, Michos ED, Kwiterovich PO, Kulkarni KR, Chimera J, Cannon CP, Blumenthal RS, Jones SR. Very large database of lipids: rationale and design. Clin Cardiol. 2013 Nov;36(11):641-8. doi: 10.1002/clc.22214. Epub 2013 Oct 1. PMID 24122913
- [Result] Martin SS, Blaha MJ, Elshazly MB, Brinton EA, Toth PP, McEvoy JW, Joshi PH, Kulkarni KR, Mize PD, Kwiterovich PO, Defilippis AP, Blumenthal RS, Jones SR. Friedewald-estimated versus directly measured low-density lipoprotein cholesterol and treatment implications. J Am Coll Cardiol. 2013 Aug 20;62(8):732-9. doi: 10.1016/j.jacc.2013.01.079. Epub 2013 Mar 21. PMID 23524048
- [Result] Ahmed, HM, Elshazly MB, Martin SS, Blaha MJ, Kulkarni KR, Jones SR. Ratio of Dense to Buoyant LDL Subclass is Associated with LDL Density Phenotype (VLDL-5). The Open Chemical and Biomedical Methods Journal 2013. 6:1-5.
- [Result] Elshazly MB, Martin SS, Blaha MJ, Joshi PH, Toth PP, McEvoy JW, Al-Hijji MA, Kulkarni KR, Kwiterovich PO, Blumenthal RS, Jones SR. Non-high-density lipoprotein cholesterol, guideline targets, and population percentiles for secondary prevention in 1.3 million adults: the VLDL-2 study (very large database of lipids). J Am Coll Cardiol. 2013 Nov 19;62(21):1960-1965. doi: 10.1016/j.jacc.2013.07.045. Epub 2013 Aug 21. PMID 23973689
- [Result] Swiger KJ, Martin SS, Blaha MJ, Toth PP, Nasir K, Michos ED, Gerstenblith G, Blumenthal RS, Jones SR. Narrowing sex differences in lipoprotein cholesterol subclasses following mid-life: the very large database of lipids (VLDL-10B). J Am Heart Assoc. 2014 Apr 22;3(2):e000851. doi: 10.1161/JAHA.114.000851. PMID 24755154
- [Result] Miller PE, Martin SS, Toth PP, Santos RD, Blaha MJ, Nasir K, Virani SS, Post WS, Blumenthal RS, Jones SR. Screening and advanced lipid phenotyping in familial hypercholesterolemia: The Very Large Database of Lipids Study-17 (VLDL-17). J Clin Lipidol. 2015 Sep-Oct;9(5):676-83. doi: 10.1016/j.jacl.2015.06.015. Epub 2015 Jul 9. PMID 26350814
- [Result] Quispe R, Manalac RJ, Faridi KF, Blaha MJ, Toth PP, Kulkarni KR, Nasir K, Virani SS, Banach M, Blumenthal RS, Martin SS, Jones SR. Relationship of the triglyceride to high-density lipoprotein cholesterol (TG/HDL-C) ratio to the remainder of the lipid profile: The Very Large Database of Lipids-4 (VLDL-4) study. Atherosclerosis. 2015 Sep;242(1):243-50. doi: 10.1016/j.atherosclerosis.2015.06.057. Epub 2015 Jul 7. PMID 26232164
- [Result] Quispe R, Al-Hijji M, Swiger KJ, Martin SS, Elshazly MB, Blaha MJ, Joshi PH, Blumenthal RS, Sniderman AD, Toth PP, Jones SR. Lipid phenotypes at the extremes of high-density lipoprotein cholesterol: The very large database of lipids-9. J Clin Lipidol. 2015 Jul-Aug;9(4):511-8.e1-5. doi: 10.1016/j.jacl.2015.05.005. Epub 2015 Jun 19. PMID 26228668
- [Result] Elshazly MB, Quispe R, Michos ED, Sniderman AD, Toth PP, Banach M, Kulkarni KR, Coresh J, Blumenthal RS, Jones SR, Martin SS. Patient-Level Discordance in Population Percentiles of the Total Cholesterol to High-Density Lipoprotein Cholesterol Ratio in Comparison With Low-Density Lipoprotein Cholesterol and Non-High-Density Lipoprotein Cholesterol: The Very Large Database of Lipids Study (VLDL-2B). Circulation. 2015 Aug 25;132(8):667-76. doi: 10.1161/CIRCULATIONAHA.115.016163. Epub 2015 Jul 2. PMID 26137953
- [Result] Lupton JR, Faridi KF, Martin SS, Sharma S, Kulkarni K, Jones SR, Michos ED. Deficient serum 25-hydroxyvitamin D is associated with an atherogenic lipid profile: The Very Large Database of Lipids (VLDL-3) study. J Clin Lipidol. 2016 Jan-Feb;10(1):72-81.e1. doi: 10.1016/j.jacl.2015.09.006. Epub 2015 Sep 25. PMID 26892123
- [Result] Lupton JR, Quispe R, Kulkarni K, Martin SS, Jones SR. Serum homocysteine is not independently associated with an atherogenic lipid profile: The Very Large Database of Lipids (VLDL-21) study. Atherosclerosis. 2016 Jun;249:59-64. doi: 10.1016/j.atherosclerosis.2016.03.031. Epub 2016 Mar 26. PMID 27065242
- [Result] Sathiyakumar V, Park J, Golozar A, Lazo M, Quispe R, Guallar E, Blumenthal RS, Jones SR, Martin SS. Fasting Versus Nonfasting and Low-Density Lipoprotein Cholesterol Accuracy. Circulation. 2018 Jan 2;137(1):10-19. doi: 10.1161/CIRCULATIONAHA.117.030677. Epub 2017 Oct 16. PMID 29038168
- [Result] Faridi KF, Lupton JR, Martin SS, Banach M, Quispe R, Kulkarni K, Jones SR, Michos ED. Vitamin D deficiency and non-lipid biomarkers of cardiovascular risk. Arch Med Sci. 2017 Jun;13(4):732-737. doi: 10.5114/aoms.2017.68237. Epub 2017 Jun 12. PMID 28721139
- [Result] Sajja A, Park J, Sathiyakumar V, Varghese B, Pallazola VA, Marvel FA, Kulkarni K, Muthukumar A, Joshi PH, Gianos E, Hirsh B, Mintz G, Goldberg A, Morris PB, Sharma G, Blumenthal RS, Michos ED, Post WS, Elshazly MB, Jones SR, Martin SS. Comparison of Methods to Estimate Low-Density Lipoprotein Cholesterol in Patients With High Triglyceride Levels. JAMA Netw Open. 2021 Oct 1;4(10):e2128817. doi: 10.1001/jamanetworkopen.2021.28817. PMID 34709388
- [Result] Chilazi M, Zheng W, Park J, Marvel FA, Khoury S, Jones SR, Martin SS. Quantifying the contribution of lipoprotein(a) to all apoB containing particles. J Clin Lipidol. 2022 Mar-Apr;16(2):220-226. doi: 10.1016/j.jacl.2022.02.004. Epub 2022 Feb 12. PMID 35241398
- [Result] Zheng W, Chilazi M, Park J, Sathiyakumar V, Donato LJ, Meeusen JW, Lazo M, Guallar E, Kulkarni KR, Jaffe AS, Santos RD, Toth PP, Jones SR, Martin SS. Assessing the Accuracy of Estimated Lipoprotein(a) Cholesterol and Lipoprotein(a)-Free Low-Density Lipoprotein Cholesterol. J Am Heart Assoc. 2022 Jan 18;11(2):e023136. doi: 10.1161/JAHA.121.023136. Epub 2022 Jan 13. PMID 35023348
- [Result] Quispe R, Brownstein AJ, Sathiyakumar V, Park J, Chang B, Sajja A, Guallar E, Lazo M, Jones SR, Martin SS. Utility of non-HDL-C and apoB targets in the context of new more aggressive lipid guidelines. Am J Prev Cardiol. 2021 May 29;7:100203. doi: 10.1016/j.ajpc.2021.100203. eCollection 2021 Sep. PMID 34611642
- [Result] Varghese B, Park J, Chew E, Sajja A, Brownstein A, Pallazola VA, Sathiyakumar V, Jones SR, Sniderman AD, Martin SS. Importance of the triglyceride level in identifying patients with a Type III Hyperlipoproteinemia phenotype using the ApoB algorithm. J Clin Lipidol. 2021 Jan-Feb;15(1):104-115.e9. doi: 10.1016/j.jacl.2020.09.011. Epub 2020 Oct 20. PMID 33189625
- [Result] Martin SS, Blaha MJ, Elshazly MB, Toth PP, Kwiterovich PO, Blumenthal RS, Jones SR. Comparison of a novel method vs the Friedewald equation for estimating low-density lipoprotein cholesterol levels from the standard lipid profile. JAMA. 2013 Nov 20;310(19):2061-8. doi: 10.1001/jama.2013.280532. PMID 24240933
- [Result] Sathiyakumar V, Pallazola VA, Park J, Vakil RM, Toth PP, Lazo-Elizondo M, Quispe R, Guallar E, Banach M, Blumenthal RS, Jones SR, Martin SS. Modern prevalence of the Fredrickson-Levy-Lees dyslipidemias: findings from the Very Large Database of Lipids and National Health and Nutrition Examination Survey. Arch Med Sci. 2019 Aug 3;16(6):1279-1287. doi: 10.5114/aoms.2019.86964. eCollection 2020. PMID 33224326
- [Result] Pallazola VA, Sathiyakumar V, Park J, Vakil RM, Toth PP, Lazo-Elizondo M, Brown E, Quispe R, Guallar E, Banach M, Blumenthal RS, Jones SR, Marais D, Soffer D, Sniderman AD, Martin SS. Modern prevalence of dysbetalipoproteinemia (Fredrickson-Levy-Lees type III hyperlipoproteinemia). Arch Med Sci. 2019 Aug 2;16(5):993-1003. doi: 10.5114/aoms.2019.86972. eCollection 2020. PMID 32863987
- [Result] Quispe R, Hendrani AD, Baradaran-Noveiry B, Martin SS, Brown E, Kulkarni KR, Banach M, Toth PP, Brinton EA, Jones SR, Joshi PH. Characterization of lipoprotein profiles in patients with hypertriglyceridemic Fredrickson-Levy and Lees dyslipidemia phenotypes: the Very Large Database of Lipids Studies 6 and 7. Arch Med Sci. 2019 Sep;15(5):1195-1202. doi: 10.5114/aoms.2019.87207. Epub 2019 Aug 22. PMID 31572464
- [Result] Faridi KF, Quispe R, Martin SS, Hendrani AD, Joshi PH, Brinton EA, Cruz DE, Banach M, Toth PP, Kulkarni K, Jones SR. Comparing different assessments of remnant lipoprotein cholesterol: The very large database of lipids. J Clin Lipidol. 2019 Jul-Aug;13(4):634-644. doi: 10.1016/j.jacl.2019.06.001. Epub 2019 Jun 11. PMID 31320236
- [Derived] Sathiyakumar V, Park J, Quispe R, Elshazly MB, Michos ED, Banach M, Toth PP, Whelton SP, Blumenthal RS, Jones SR, Martin SS. Impact of Novel Low-Density Lipoprotein-Cholesterol Assessment on the Utility of Secondary Non-High-Density Lipoprotein-C and Apolipoprotein B Targets in Selected Worldwide Dyslipidemia Guidelines. Circulation. 2018 Jul 17;138(3):244-254. doi: 10.1161/CIRCULATIONAHA.117.032463. Epub 2018 Mar 5. PMID 29506984
- See also: Very Large Database of Lipids — https://clinicaltrials.gov/study/NCT07169266?limit=10&sort=@relevance&term=%09NCT07169266&rank=1